CLINICAL TRIAL: NCT05518721
Title: Synthetic Cartilage Implant Versus Interposition Arthroplasty in Hallux Rigidus Treatment: A Randomized Clinical Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Original PI left institution and successor has no interest in continuing project.
Sponsor: John Femino (Other)
Responsible Party: Sponsor-Investigator, John Femino, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202010411
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Hallux Rigidus
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Synthetic Cartilage Implant (Active Comparator)
  Interventions: Procedure: Hallux Rigidus Treatment
- Dermal Interposition Arthroplasty (Active Comparator)
  Interventions: Procedure: Hallux Rigidus Treatment

INTERVENTIONS:
Procedure: Hallux Rigidus Treatment — Participants will receive either a synthetic cartilage implant or dermal interposition arthroplasty

SUMMARY:
A minimum of 100 patients with grade III hallux rigidus will be randomized in two parallel groups for surgical care. The first group will be submitted to the insertion of a synthetic cartilage implant at the metatarsophalangeal (MTP) joint. The second group will receive a dermal interposition arthroplasty at the MTP. Both sides will undergo the same post-operative protocol. Pain, complications, and functional results will be evaluated in a minimal of two years of follow-up.

DETAILED DESCRIPTION:
A minimum of 100 patients with grade III hallux rigidus will be randomized in two parallel groups for surgical care. The first group will be submitted to the insertion of a synthetic cartilage implant at the metatarsophalangeal (MTP) joint. The second group will receive a dermal interposition arthroplasty at the MTP. Both sides will undergo the same post-operative protocol. Pain, complications, and functional results will be evaluated in a minimal of two years of follow-up.

The synthetic implant begins by performing and dorsal midline approach, from the proximal phalanx diaphysis to the first metatarsal neck. Dissection is carried avoiding injury to the dorsal cutaneous nerves and the extensor hallucis longus tendon. The capsule is open longitudinally, osteophytes removed, and a guidewire inserted through the center of the first metatarsal head. The position of the metallic wire is checked and the tunnel for the implant is drilled. The synthetic cartilage implant (Cartiva™, Stryker Medical®) is introduced through the tunnel, leaving it proud with the head surface by 2mm. The capsule is closed, followed by the other planes and the skin. The patient is banded and placed in a postoperative hard sole shoe for six weeks. Range of motion is encouraged from the third week and the shoe is discontinued after the sixth week. Return to sports activities and normal shoewear occurs by twelve weeks.

The interposition arthroplasty initiates with the same dorsal midline approach, from the proximal phalanx diaphysis to the first metatarsal neck. Dissection is carried avoiding injury to the dorsal cutaneous nerves and the extensor hallucis longus tendon. The capsule is open longitudinally and osteophytes are removed. A guidewire inserted through the center of the first metatarsal head and the center of the proximal phalanx for proper surface preparation. Convex-concaves anatomical drills are used, removing remaining cartilage and opening space for the graft. A decellularized dermal allograft (Arthroflex™, Arthrex®) is placed at the joint and sutured to the head, maintaining the epidermal surface in contact with the phalanx. The graft is trimmed, the capsule is closed, which is followed by the other planes and the skin. The patient is banded and placed in a postoperative hard sole shoe for six weeks. Range of motion is encouraged from the third week and the shoe is discontinued after the sixth week. Return to sports activities and normal shoewear occurs by twelve weeks.

The WBCT is the standard of care for the preoperative and postoperative assessment of patients with hallux rigidus. Some of the complications will also be evaluated through WBCT. No extra WBCT will be performed other than what we normally do for patients.

Randomization will be performed previously at the beginning of the study and will be performed by an outside researcher. Allocation will happen during surgery scheduling.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be older than 18 and younger than 75 years of age, both genders.
* Participants must be experiencing symptoms related to their baseline condition for at least six months before the surgery.
* Clinical and radiographical clinical diagnosis of hallux rigidus.
* Hallux Rigidus grade III or grade IV.
* Surgical indication after failure of nonoperative treatment (at least six months).

Exclusion Criteria:

* Previous hallux metatarsophalangeal fusion.
* Less than 20 degrees of complete range of motion on the hallux metatarsophalangeal joint.
* Patient desire or medical indication for a hallux metatarsophalangeal joint arthrodesis.
* Patient desire or medical indication for other surgical modalities.
* History or documented evidence of autoimmune or peripheral vascular diseases.
* History or documented evidence of peripheral neuropathy (nervous compression syndrome, tarsal tunnel syndrome) or systemic inflammatory disease a (rheumatoid arthritis, seronegative, connective, etc.).
* Any condition that represents a contraindication of the proposed therapies.
* Any physical or social limitation that makes the protocol continuation unviable.
* Impossibility or incapacity to sign the informed Consent Form.
* Presence of infectious process (superficial on the skin and cellular tissue, or deep in the bone) in the region to be treated.
* Pregnancy.
* Clinical and imaging diagnosis of untreated osteoporosis.
* Serum vitamin D levels below 20ng/ml.
* Non-palpable anterior or posterior tibial pulse; or abnormal capillary filling.
* Tumor lesions (primary or secondary tumors).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-05 (Estimated); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes | 96 weeks post-surgery
  To compare patient reported outcomes (PROs) of patients undergoing HR treatment using a synthetic implant and utilizing interposition arthroplasty.

SECONDARY OUTCOMES:
Survival | 6 months post-surgery
  To compare survival rate (reoperation) between the two techniques.
Complications | 6 months post-surgery
  To compare major and minor complications between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: John Femino, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No